CLINICAL TRIAL: NCT04096612
Title: The Therapeutic Effect of Dysthyroid Optic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: yanghs2018
Record Dates: First submitted 2018-12-27; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orbital decompression combined MPT (Experimental): Orbital decompression was performed by the same doctor with rich clinical experience. MPT should be implemented in the patients with obvious thyroid disorder before orbital decompression surgery which should only be performed when thyroid function was stabilized. The surgery was performed under general anesthesia. An arcuate incision was made in the skin 2 mm below the lower eyelid margin, and the tissue under the incision were separated to the periorbita and orbital septum. Part of the medial orbital wall, inferior orbital wall and partial tissue of ethmoidal sinus were removed, and an appropriate amount of adipose tissue was excised. MPT was conducted after the surgery, at a dose of 1g methylprednisolone per day through intravenous injection for 3 consecutive days with a total amount of 3g methylprednisolone. After 3 days of intravenous injection of methylprednisolone, prednisone was orally taken by the patients at a dose of 30 mg/day which was gradually reduced.
  Interventions: Procedure: Orbital decompression combined with MPT
- Separate MPT (Experimental): MPT was conducted after the surgery, at a dose of 1g methylprednisolone per day through intravenous injection for 3 consecutive days with a total amount of 3g methylprednisolone. After 3 days of intravenous injection of methylprednisolone, prednisone was orally taken by the patients at a dose of 30 mg/day which was gradually reduced.
  Interventions: Procedure: Orbital decompression combined with MPT

INTERVENTIONS:
Procedure: Orbital decompression combined with MPT — Orbital decompression combined with MPT

SUMMARY:
Thyroid associated ophthalmopathy (TAO) is a common autoimmune disorder. The pathogenesis of TAO is unclear, and studies found that T cell, B cell and monocytes, macrophages and mast cells are located in the orbital tissue of TAO. Dysthyroid optic neuropathy (DON) is the most serious complication of TAO, which can cause blurred vision, color vision and vision function damage, and affects the quality of life. Investigation of the therapeutic effect of orbital decompression may provide some clues to make the policy at treatment of DON. We explore the therapeutic effect of orbital decompression in patients with DON in both eyes.

ELIGIBILITY:
Inclusion Criteria:

- Ability to perform visual fields and VEP examination Without any serious systemic diseases Without any surgery on eyes in six months

Exclusion Criteria:

- With any serious systemic diseases With any surgery on eyes in six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
BCVA | 6 months
  best corrected visual acuity in logMAR
IOP | 6 months
  intraocular pressure in mmHg
proptosis | 6 months
  proptosis in mm
upper eyelid retraction | 6 months
  upper eyelid retraction in mm
CAS | 6 months
  clinical activity score

SECONDARY OUTCOMES:
MD | 6 months
  mean deviation of visual field in dB
PSD | 6 months
  pattern standard deviation of visual field in dB

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol